CLINICAL TRIAL: NCT00395694
Title: Clinical Evaluation of BW430C in Epilepsy<Phase III Study>
Brief Title: Clinical Evaluation of BW430C in Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM107844
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: epilepsy; Incidence of rash; safety evaluation for initial dose; patients with Valproic acid
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

ARMS (1):
- lamictal (Experimental)
  Interventions: Drug: lamictal

INTERVENTIONS:
Drug: lamictal — anti-epileptic drug

SUMMARY:
To evaluate safety information of BW430C when administered using the lower starting doses and slower dose escalations as recommended Global Data Sheet

ELIGIBILITY:
Inclusion criteria:

* Epilepsy with partial seizures
* Tonic clonic seizures
* Generalized seizures of Lennox-Gastaut
* Subjects whose seizures are easily recognizable at least one seizure per month and counts for 8 consecutive weeks prior to the start of the study drug.
* Concurrent AEDs: Subjects taking concurrent VPA.

Exclusion criteria:

* Previous participation in a study of Lamictal
* Known hypersensitivity to any drugs
* Pregnant women
* nursing mothers
* women who may be pregnant
* women contemplating pregnancy during the study period

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-08-07; Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Kumamoto, Japan
- GSK Investigational Site

REFERENCES:
- [Background] Shunsuke Ohtahara, Tateki Fujiwara, Sunao Kaneko, Masafumi Iijima. Clinical Evaluation of Lamotrigine with the Current Recommended Dose in Overseas - Phase III study of lamotrigine in patients with epilepsy treated with valproate - . [J.New Rem. & Clin. Vol.57 No.9 2008]. 2008;57(J.New Rem. & Clin):1442-1453.

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults: LTG: Adult participants were initiated on 12.5 milligrams per day (mg/day) of BW430C (lamotrigine [LTG]) (as a tablet taken orally) once daily. Participants had their dose increased to an optimal maintenance dose (escalation phase) and then were maintained at that dose for 8 weeks (maintenance phase [MP]). During the 8-week MP, participants received up to a maximum of 200 mg/day for adults taking valproeic acid (VPA) or up to a maximum of 400 mg/day for adults not taking VPA plus an inducer of LTG glucuronidation. Participants who achieved adequate seizure control at the end of the MP and for whom no alternative antiepileptic drugs (AEDs) were available were allowed to continue treatment with LTG until the drug is marketed (continuation phase).
- Adolescents: LTG: Adolescent participants were initiated on 0.15 mg/kilogram (kg)/day. Participants had their dose increased to an optimal maintenance dose (escalation phase) and then were maintained at that dose for 8 weeks (MP). During the 8-week MP, adolescents taking VPA alone received up to a maximum of 3 mg/kg/day, adolescents taking VPA with an inducer of LTG glucuronidation received up to a maximum of 5 mg/kg/day, and adolescents not taking VPA with an inducer of LTG glucuronidation received up to a maximum of 15 mg/kg/day. Participants who achieved adequate seizure control at the end of the MP and for whom no alternative AEDs were available were allowed to continue treatment with BW430C until the drug is marketed (continuation phase).
Period: Escalation Phase + Maintenance Phase
Arm/Group | Adults: LTG | Adolescents: LTG
Started | 51 | 51
Completed | 50 | 49
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2
Period: Continuation Phase
Arm/Group | Adults: LTG | Adolescents: LTG
Started | 49 (One participant completing the Escalation/Maintenance Phase did not start the Continuation Phase.) | 48 (One participant completing the Escalation/Maintenance Phase did not start the Continuation Phase.)
Completed | 34 | 35
Not Completed | 15 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 12 | 11
Not completed — Withdrawal Due to Wishes of Family | 1 | 0
Not completed — Poor Compliance | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults: LTG | Adolescents: LTG | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (9.9) | 8.2 (4.1) | 18.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 28 | 26 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Rash Event (Including Stevens-Johnson Syndrome [SJS] and Any Other Serious Drug Eruption) During the Initial 8 Weeks of Study Treatment
Description: Any rash event (including SJS or any other serious drug eruption) includes: all event terms containing "rash"; drug eruption; SJS; toxic epidermal necrolysis; rash generalized; and events grouped into the "Skin and Subcutaneous Tissue Disorders" system organ class per the Medical Dictionary for Regulatory Activities (MedDRA), including the above-mentioned events that the GSK medical advisors judged to be included as any rash event. SJS, also called as erythema multiforme, is a skin disorder resulting from an allergic reaction or infection.
Time Frame: 8 weeks
Population: Safety Population: all participants enrolled in the study who received at least one dose of study medication
Measure: Number; unit: participants
Groups:
- Total: LTG: Adult participants were initiated on 12.5 mg/day, and adolescents were initiated on 0.15 mg/kg/day. Participants had their dose increased to an optimal maintenance dose (escalation phase) and then were maintained at that dose for 8 weeks (MP). During the 8-week MP, participants received up to a maximum of 200 mg/day for adults taking VPA or up to a maximum of 400 mg/day for adults not taking VPA plus an inducer of LTG glucuronidation. During the MP, adolescents taking VPA alone received up to a maximum of 3 mg/kg/day, adolescents taking VPA with an inducer of LTG glucuronidation received up to a maximum of 5 mg/kg/day, and adolescents not taking VPA with an inducer of LTG glucuronidation received up to a maximum of 15 mg/kg/day. Participants who achieved adequate seizure control at the end of the MP and for whom no alternative AEDs were available were allowed to continue treatment with BW430C until the drug is marketed (continuation phase).
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 51 | 51 | 102
participants | 2 | 3 | 5
Statistical Analysis 1: Comparison: Total: LTG; Test type: Superiority or Other; Percentage of participants = 4.9, 95% CI 2-sided [1.6 to 11.1] — The estimated value represents the percentage of participants with rash events

2. Secondary Outcome: Number of Rash Events Experienced (Including SJS and Any Other Serious Drug Eruption) During the Initial 8 Weeks of Study Treatment
Description: as for outcome 1
Time Frame: 8 weeks
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: rash events
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 2 | 3 | 5
rash events | 3 | 4 | 7

3. Secondary Outcome: Number of Participants With the Indicated Intensity of Rash (Including SJS and Any Other Serious Drug Eruption) During the Initial 8 Weeks of Study Treatment
Description: The rash events (including SJS and any other serious drug eruption) were classified into severe (rash prevents participant from leading a normal life), moderate (participant's discomfort due to rash interferes with daily life), and mild (no interference with participant's daily life due to rash), based on the intesity of the event.
Time Frame: 8 weeks
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: participants
Arm/Group | Total: LTG
Number analyzed (Participants) | 5
participants
  Severe | 0
  Moderate | 2
  Mild | 3

4. Secondary Outcome: Number of Drug-related and Not Related Rash Events (Including SJS and Any Other Serious Drug Eruption) During the Initial 8 Weeks of Study Treatment
Description: The adverse event of rash was considered to be drug-related when the Investigator answered "Yes" to the following question: "Is there a reasonable possibility that the adverse event may have been caused by the investigational product?".
Time Frame: 8 weeks
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: rash events
Arm/Group | Total: LTG
Number analyzed (Participants) | 5
rash events
  Drug related | 3
  Not related to drug | 4

5. Secondary Outcome: Percentage of Participants With at Least a 50 Percent Reduction in Seizure Frequency for the Indicated Types of Seizures
Description: Partial seizures are seizures that affect only a part of the brain at onset. Tonic-clonic seizures (grand mal seizures) affect the entire brain and are characterized by a generalized involuntary muscular contraction and cessation of respiration followed by tonic and clonic spasms of the muscles. Lennox-Gastaut syndrome (LGS) is a pediatric epilepsy syndrome characterized by multiple seizure types; mental retardation or regression; and abnormal findings on an electroencephalogram (EEG), with paroxysms of fast activity and generalized slow spike-and-wave discharges.
Time Frame: 8 weeks
Population: Full Analysis Set (FAS) Population: all enrolled participants except those who had no assessments of the main efficacy variable (percent reduction in seizure frequency).
Measure: Number; unit: percentage of participants
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 28 | 25 | 53
percentage of participants
  All Partial Seizures, n=28, 25, 53 | 17.9 | 20.0 | 18.9
  Tonic-clonic Seizures, n=5, 4, 9 | 60.0 | 0 | 33.3
  Generalized Seizures with LGS, n=25, 25, 50 | 16.0 | 20.0 | 18.0

6. Secondary Outcome: Percent Change in Seizure Frequency of the Indicated Types of Seizures
Description: Percent change in seizure frequency was calculated as 100 * (pre-treatment seizures minus MP seizures)/pre-treatment seizures. Partial seizures are seizures that affect only a part of the brain at onset. Tonic-clonic seizures (grand mal seizures) affect the entire brain and are characterized by a generalized involuntary muscular contraction and cessation of respiration followed by tonic and clonic spasms of the muscles. Lennox-Gastaut syndrome (LGS) is a pediatric epilepsy syndrome characterized by multiple seizure types, mental retardation or regression, and abnormal findings on an ECG.
Time Frame: Pre-treatment (Day 0) and Week 8 of the Maintenance Phase (Study Week 14)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 28 | 25 | 53
percent change
  All Partial Seizures, n=28, 25, 53 | 6.3 [-44.8 to 28.7] | -11.1 [-46.6 to 34.6] | -9.8 [-42.3 to 28.6]
  Tonic-clonic Seizures, n=5, 4, 9 | 83.3 [NA to NA] — The 95% confidence interval cannot be calculated because fewer than 10 events occurred. | 27.4 [NA to NA] — The 95% confidence interval cannot be calculated because fewer than 10 events occurred. | 36.5 [-47.9 to 100.0]
  Generalized Seizures with LGS, n=25, 25, 50 | 18.6 [-16.2 to 32.2] | 10.1 [-24.9 to 28.8] | 12.4 [5.8 to 27.6]

7. Secondary Outcome: Number of Participants With Any Rash Event (Including SJS and Any Other Serious Drug Eruption) up to the End of the Maintenance Phase
Description: as for outcome 1
Time Frame: Up to Week 8 of the Maintenance Phase (Study Week 14)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 51 | 51 | 102
participants | 2 | 3 | 5

8. Secondary Outcome: Number of Rash Events Experienced (Including SJS and Any Other Serious Drug Eruption) up to the End of the Maintenance Phase
Description: as for outcome 1
Time Frame: Up to Week 8 of the Maintenance Phase (Study Week 14)
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: rash events
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 2 | 3 | 5
rash events | 3 | 4 | 7

9. Secondary Outcome: Number of Participants With the Indicated Intensity of Rash (Including SJS and Any Other Serious Drug Eruption) up to the End of the Maintenance Phase
Description: as for outcome 3
Time Frame: Up to Week 8 of the Maintenance Phase (Study Week 14)
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: participants
Arm/Group | Total: LTG
Number analyzed (Participants) | 5
participants
  Severe | 0
  Moderate | 2
  Mild | 3

10. Secondary Outcome: Number of Drug-related and Not Related Rash Events (Including SJS and Any Other Serious Drug Eruption) up to the End of the Maintenance Phase
Description: as for outcome 4
Time Frame: Up to Week 8 of the Maintenance Phase (Study Week 14)
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: rash events
Arm/Group | Total: LTG
Number analyzed (Participants) | 5
rash events
  Drug related | 3
  Not related to drug | 4

11. Secondary Outcome: Number of Rash Events (Including SJS and Any Other Serious Drug Eruption) Adjudicated by the Rash Adjudication Committee in Participants Taking VPA
Description: The rash adjudication committee reviewed all rash events from a dermatologic standpoint based on the nature, onset site, affected area, time to onset, outcome, and the investigator's comments to adjudicate whether or not the reported event was a drug eruption. A drug eruption is an eruption or a solitary lesion caused by a drug taken internally, often a result of allergic sensitization.
Time Frame: Up to Week 8 of the Maintenance Phase (Study Week 14)
Population: Safety Population. Only those participants who had experienced any rash event were evaluated.
Measure: Number; unit: adjudicated rash events
Units Other Than Participants: total rash events
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Number analyzed (Participants) | 2 | 3 | 5
Number analyzed (total rash events) | 3 | 4 | 7
adjudicated rash events | 1 | 2 | 3

12. Secondary Outcome: Percentage of Participants With Monocyte Values Outside the Normal Range (Shifted High) at Weeks 4 and 8
Description: Monocytes are a type of white blood cell (WBC; typically comprising 2%-8% of total WBCs) and are a part of the immune system. The normal range for adults is 0.2 to 0.95 * 10^3 cells per microliter (µL); the normal range for adolescents is 0 to 0.8 * 10^3 cells per µL. The monocyte count may increase during chronic inflammation, stress response, immune-mediated disease, viral fever, etc. The percentage of participants (par.) with monocyte values outside the normal range was calculated as 100 * (number of par. with monocyte values outside the normal range) divided by the total number of par.
Time Frame: Week 4 and Week 8
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Total: LTG
Number analyzed (Participants) | 102
percentage of participants
  Week 4 | 15.2
  Week 8 | 16.2

ADVERSE EVENTS:
Arm/Group | Adults: LTG | Adolescents: LTG | Total: LTG
Serious Adverse Events (participants affected / at risk) | 5/51 | 2/51 | 7/102
Other Adverse Events (participants affected / at risk) | 48/51 | 50/51 | 98/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults: LTG (N=51) | Adolescents: LTG (N=51) | Total: LTG (N=102)
Sleepiness (Nervous system disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Aleviatin (phenytoin) poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Frequent convulsions (Nervous system disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adults: LTG (N=51) | Adolescents: LTG (N=51) | Total: LTG (N=102)
Nasopharyngitis (Infections and infestations) | 10 | 14 | 24
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 15 | 20
Somnolence (Nervous system disorders) | 7 | 11 | 18
Diarrhoea (Gastrointestinal disorders) | 3 | 11 | 14
Pyrexia (General disorders) | 7 | 6 | 13
Contusion (Injury, poisoning and procedural complications) | 8 | 4 | 12
Dizziness (Nervous system disorders) | 10 | 2 | 12
Vomiting (Gastrointestinal disorders) | 4 | 7 | 11
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 9 | 10
Excoriation (Injury, poisoning and procedural complications) | 6 | 2 | 8
Erythema (Skin and subcutaneous tissue disorders) | 1 | 6 | 7
Constipation (Gastrointestinal disorders) | 3 | 4 | 7
Pharyngitis (Infections and infestations) | 3 | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Affect lability (Psychiatric disorders) | 1 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.